CLINICAL TRIAL: NCT05085041
Title: Effectiveness of Multi-Component eHealth Intervention, Namely Healthy Online Parental Education (HOPE), to Increase Fruit and Vegetable Consumption and Active Playtime Among Toddlers at Home
Brief Title: Healthy Online Parental Education Project to Increase Fruit and Vegetable Intake and Active Playtime Among Toddlers
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB2021-505
Record Dates: First submitted 2021-09-13; First posted 2021-10-20 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Eating Behavior
Keywords: Child Nutrition; Carotenoid Levels; Obesity; Feeding Practice; Child and Maternal Nutrition; Screen Time; Mixed-Methods Research
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: This research project will include two groups; the intervention and the control groups. Participants will be randomly assigned via block randomization with selected block sizes of 4. Randomization will be conducted by a researcher not involved in data management. The statistical software R version 3.5.1 will be used to determine to generate randomized arm allocation sequences through a fixed seed. The randomization will be stratified by centers. Those allocation sequences will be printed out and individually stored in serially numbered, opaque, sealed envelopes. Participants will be informed of group allocation via opaque and sealed envelopes after the collection of baseline data. Participants in the intervention group will receive 8 sessions of an online multi-component nutrition intervention. The control group will receive a copy of the booklet that includes dietary recommendations for adults and children, followed by the 2020 U.S. Department of Agriculture Dietary Guidelines.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The participants in this group will receive 8 sessions of a multi-component online education intervention. The education curriculum will be focused on addressing evidence-based healthy habits that are related to preventing childhood obesity: more vegetables and fruits, less screen time, and more physical activity. Topics may include age-appropriate nutrition and eating, picky eating, positive parental feeding practices, active playtime, and screen time. Strategies for eating healthy on a budget will be also provided to the participants.
  The intervention will incorporate multi-component as follow: instructional YouTube videos, online cooking activities, reminder text messages with key information, and telephone consultation. Each session will include a lifestyle component regarding eating, feeding, and physical activity, aimed at equipping parents with knowledge and skills to improve fruit and vegetable intake and physical activity levels of young children.
  Interventions: Behavioral: Multi-Component eHealth Intervention, namely Healthy Online Parental Education (HOPE)
- Control Group (No Intervention): The participants in the control group will receive no intervention. However, the investigators will provide the control group with a copy of the booklet that includes 2020 USDA dietary guidelines for a healthy diet for young children. This will enable the investigators to see if the multi-component education intervention (stated above) is more effective on behavior changes than the written booklet in the control group.

INTERVENTIONS:
Behavioral: Multi-Component eHealth Intervention, namely Healthy Online Parental Education (HOPE) — The investigators will provide 8 sessions of a multi-component education intervention to the participants in the intervention group. Each session will address parental nutrition knowledge, self-efficacy, and attitudes around feeding, parental modeling of healthy foods, and skill development to increase success in making behavioral changes. The intervention curriculum will be informed by Social Cognitive Theory to help parents guide young children to engage in healthy eating behaviors through modeling (Curriculum Design). The investigators will deliver the intervention using multicomponent to enhance and maximize the learning experiences of the participants for successful behavior changes. The intervention will be comprised of instructional videos, text messages with key information, online cooking activities, and telephone consultation (Modality).
  Other Names: HOPE
  Arms: Intervention Group

SUMMARY:
The research proposal will be an 8-week randomized control trial (RCT) to examine the efficacy of an eHealth intervention, namely Healthy Parental Online Education (HOPE), on fruit and vegetable intake and active playtime among toddlers enrolled in early head start programs in Lubbock, Texas. Parents with toddlers ages one to three years will be recruited from Early Head Start centers. Written consent forms will be obtained before baseline data collection. The participants will be then randomly assigned to the intervention or control group. The participants in the intervention group will receive a multi-component online nutrition intervention for eight weeks. While the control group will receive a copy of the booklet that includes the 2020 U.S. Department of Agriculture Dietary Guidelines (USDA) for toddlers and adults.

The investigators will measure sociodemographic, parental nutritional knowledge, parental attitude related to healthy eating, parental self-efficacy, parental feeding practices, carotenoids in the skin of both parents and toddlers, three-day food photos, and physical activity and sedentary times of toddlers. This research proposal hypothesizes that there will be significant differences in fruit and vegetable intake and physically active time among toddlers between the intervention and control group from baseline to 3 months. The investigators also hypothesize that there will be significant differences in parental nutrition knowledge, attitude, self-efficacy, and feeding practice between the intervention and control group from baseline to 3 months.

DETAILED DESCRIPTION:
The investigators will examine the efficacy of an eHealth intervention, namely Healthy Parental Online Education (HOPE), to increase fruit and vegetable intake and active playtime among toddlers enrolled in Early Head Start programs in Lubbock. This study will be an 8-week randomized control trial (RCT). Participants will be randomly assigned to the intervention or control group via block randomization with randomly selected block sizes of 4. Randomization will be conducted by a researcher not involved in data management. The statistical software R version 3.5.1 will be used to determine to generate randomized arm allocation sequences through a fixed seed. The randomization will be stratified by centers. Those allocation sequences will be printed out and individually stored in serially numbered, opaque, sealed envelopes. Participants will be informed of group allocation via opaque and sealed envelopes after the collection of baseline data.

Participants in the intervention group will receive 8 sessions of online multi-component HOPE nutrition intervention. While the control group will receive no intervention, the investigators will provide the control group with a copy of the booklet. This booklet will include basic nutrition recommendations for a healthy diet for adults and children, consistent with 2020 U.S. Department of Agriculture dietary guidelines.

Pre- and post-assessment will be conducted to see changes in variables of interest from baseline (T1), post-intervention (T2), to 3 months (T3). Sociodemographic and anthropometrics of parents and toddlers will be measured at T1. The investigators will also measure carotenoids in the skin of both parents and children using the Veggie Meter (Longevity Link, Salt Lake City, UT) to assess fruit and vegetable intake. Parental nutritional knowledge, attitudes related to healthy eating and activity, feeding practices, and self-efficacy will be assessed using a self-administered questionnaire. The research team will also ask parents to recall the physical activity and sedentary times of toddlers using a self-report survey. Parents will take electronic food photos using their mobile devices for three days to capture the food and beverage intake of toddlers at home. The same measurements and survey will be used at T2 except for variables related to anthropometrics and sociodemographics. Finally, the investigators will only measure the food intake of toddlers, physically active and sedentary times of toddlers, and carotenoid levels of parents and toddlers at T3, using the same methods and procedures mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Having a child between 12 and 36 months of age
* Physically and mentally capable of communicating, reading, and writing in English
* An informed consent form obtained
* Willing and able to attend the intervention

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Changes in Fruit and Vegetable Intake (Unit: Servings) | Changes in Fruit and Vegetable Intakes by toddlers from baseline to 3 months
  The investigators will assess changes in fruit and vegetable intakes by toddlers. Electronic photos will be used by parents to record food intake of toddlers. The investigators will manually count and categorize the servings of fruits and vegetables from the food photos.
Changes in Skin Carotenoid Score (Unit: nm) | Changes in Skin Carotenoid Scores by parents and toddlers from baseline to 3 months
  The Veggie Meter uses reflection spectroscopy and is an objective, noninvasive measure of the level of carotenoid pigments in a person's skin. Fruits and vegetable intakes as reflected in skin carotenoid scores will be measured by parents and toddlers, using the Veggie Meter.
Changes in Times Being Physically Active (Unit: Minutes) | Changes in Times Being Physically Active by toddlers from baseline to 3 months
  Parents will be asked to report the frequency and duration of different moderate-to-vigorous physical activity (MVPA) and sedentary activities (SA) in which toddlers were engaged during the past weekend at home. The investigators will use a proxy-reported questionnaire to capture and estimate daily minutes of MVPA and SA.

SECONDARY OUTCOMES:
Changes in Parental Nutritional Knowledge Score (Unit: Numerical Score) | Changes in Parental Nutritional Knowledge Scores from baseline to 3 months
  The investigators will use a multiple-choice questionnaire to test if there is any change in parental nutritional knowledge after the intervention.
Changes in Parental Attitude Score (Unit: Numerical Score) | Changes in Parental Attitudes Scores from baseline to 3 months
  A 13-item, responding to a 5-point Likert scale, will be assessed parental attitudes towards healthy eating and physical activity.
Changes in Parental Self-Efficacy Score (Unit: Numerical Score) | Changes in Parental Self-Efficacy Scores from baseline to 3 months
  The self-efficacy questionnaire, consisting of 8 items, will be used to assess parental self-efficacy in feeding toddlers and mealtime interaction.
Changes in Parental Feeding Practices (Unit: Numerical Score) | Changes in Parental Feeding Practices Scores from baseline to 3 months
  The Comprehensive Feeding Practices Questionnaire (CFPQ) will be used to capture a broad range of parental feeding practices and behaviors. The investigators will assess if there was any change in positive or negative feeding practices among the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Wilna Oldewage-Theron, PhD, Study Chair — Texas Tech University; Hyunjung Lee, MS, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University Center for Early Head Start, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with an academic interest in community nutrition. Data shared will be coded with no Protected Health Information (PHI) included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with requesting party.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to Individual Participant Data (IPD) can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal, statistical plan (SAP), and analytic code. For more information or to submit a request, please contact wilna.oldewage@ttu.edu.